CLINICAL TRIAL: NCT02202759
Title: A Phase 2 Trial of MLN0264 in Previously Treated Patients With Metastatic or Recurrent Adenocarcinoma of the Stomach or Gastroesophageal Junction Expressing Guanylyl Cyclase C (GCC)
Brief Title: A Study of MLN0264 in Participants With Cancer of the Stomach or Gastroesophageal Junction
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Business Decision, No Safety or Efficacy Concerns
Sponsor: Millennium Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: C26002; U1111-1155-9023 (Other: WHO); 2014-000804-88 (EudraCT Number); REec-2014-1176 (Registry Identifier: REec)
Record Dates: First submitted 2014-07-07; First posted 2014-07-29 (Estimated); Results first posted 2017-05-15 (Actual); Last update posted 2017-05-15 (Actual); Status verified 2017-04

CONDITIONS: Adenocarcinoma of the Stomach; Gastroesophageal Junction Expressing Guanylyl Cyclase C
Keywords: Drug therapy
MeSH Terms: interventions — indusatumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- MLN0264 1.8 mg/kg (Experimental): MLN0264 1.8 mg/kg, 30-minute intravenous (IV) infusion, Day 1 of each 21-day cycle, for up to 1 year or until disease progression or unacceptable toxicity occurs (Up to 14 cycles). The dose may be decreased, delayed or discontinued in participants who develop treatment-associated nonhematologic and hematologic toxicity to MLN0264.
  Interventions: Drug: MLN0264

INTERVENTIONS:
Drug: MLN0264 — MLN0264 IV infusion

SUMMARY:
The purpose of this study is to assess the efficacy, safety and tolerability of MLN0264 in patients with recurrent or metastatic guanylyl cyclase C (GCC)-positive adenocarcinoma of the stomach or gastroesophageal junction.

DETAILED DESCRIPTION:
The drug being tested in this study is called MLN0264. MLN0264 is being tested to treat tumors in people who have metastatic or recurrent gastric or gastroesophageal junction malignancies expressing guanylyl cyclase C (GCC). Participants will be analyzed in cohorts based on GCC expression: low=combined H-score 10-109, intermediate=combined H-score 110-249, high=combined IHC H-score >250. This study will assess tumor size reduction in patients who are administered MLN0264.

The study enrolled 38 patients. All participants will be administered MLN0264 at 1.8 mg/kg as a single, 30-minute, intravenous (IV) infusion on Day 1 of each 3-week treatment cycle, followed by a rest period of 20 days. Participants will continue to receive MLN0264 for up to 1 year or until disease progression or unacceptable toxicity occurs.

This multi-centre trial will be conducted worldwide. The overall time to participate in this study is approximately 19 months. Participants will make 3 to 6 visits to the clinic per treatment cycle, an end-of-treatment visit 30 days after the last dose of study medication, and follow-up assessments every 12 weeks until death or 6 months after the last patient completes treatment - whichever occurs first.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female participants 18 years of age or older when written informed consent is obtained.
2. Histologically confirmed metastatic or advanced inoperable adenocarcinoma of the stomach or gastroesophageal junction with immunohistochemistry (IHC) evidence of guanylyl cyclase C (GCC) expression indicated by an H-score of 10 or greater.
3. Treatment with 1 or more prior chemotherapies for advanced or metastatic adenocarcinoma of the stomach or gastroesophageal junction.
4. Measurable disease as defined by Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1 guidelines. All scans and x-rays used to document measurable disease must be done within 28 days before enrollment (ascites and bone lesions are not considered measureable disease).
5. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1 within 14 days before enrollment.
6. Female participants who:

   * Are postmenopausal for at least 1 year before the screening visit, OR
   * Are surgically sterile, OR
   * If they are of childbearing potential, agree to practice 2 effective methods of contraception, at the same time, from the time of signing the informed consent through 30 days after the last dose of study drug, or
   * Agree to practice true abstinence, when this is in line with the preferred and usual lifestyle of the participant. (Periodic abstinence [eg, calendar, ovulation, symptothermal, postovulation methods] and withdrawal are not acceptable methods of contraception.)

   Male participants, even if surgically sterilized (ie, status postvasectomy), who:
   * Agree to practice effective barrier contraception during the entire study treatment period and through 4 months after the last dose of study drug, or
   * Agree to practice true abstinence, when this is in line with the preferred and usual lifestyle of the participant. (Periodic abstinence [eg, calendar, ovulation, symptothermal, postovulation methods for the female partner] and withdrawal are not acceptable methods of contraception.)
7. Voluntary written consent must be given before performance of any study-related procedure not part of standard medical care, with the understanding that consent may be withdrawn by the participant at any time without prejudice to future medical care.
8. Adequate organ and hematological function as evidenced by the following laboratory values within 14 days before enrollment:

   * Absolute neutrophil count (ANC) ≥ 1.5 x 10^9/L
   * Platelet count ≥ 100 x 10^9/L
   * Hemoglobin ≥ 9 g/dL
   * Activated partial thromboplastin time (aPTT) ≤ 1.5 x the upper limit of the normal range (ULN) per institutional laboratory normal range
   * International normalized ratio (INR) ≤ 1.5 x ULN
   * Serum creatinine ≤ 1.5 x ULN
   * Total bilirubin ≤ 1.5 x ULN
   * Albumin ≥ 3g/dL
   * Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 2.5 x ULN
   * Serum lipase ≤ 3 x ULN and serum amylase within the normal range
9. Resolution of all toxic effects of prior treatments except alopecia to Grade 0 or 1 by National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) version 4.03.
10. Willing and able to comply with scheduled visits, treatment plan, laboratory tests, and other trial procedures.

Exclusion Criteria:

1. Radiotherapy within 4 weeks before enrollment.
2. Concurrent treatment or treatment within 4 weeks of study entry with any other investigational agent or chemotherapy.
3. Female participants who are lactating and breastfeeding or have a positive pregnancy test during the Screening period.
4. Uncontrolled, clinically significant, symptomatic cardiovascular disease within 6 months before enrollment, including myocardial infarction, unstable angina, Grade 2 or greater peripheral vascular disease, cerebrovascular accident, transient ischemic attack, congestive heart failure, or arrhythmias not controlled by outpatient medication.
5. Treatment with any medication that has a clinically relevant potential risk of prolonging the QT interval or inducing torsades de pointes that cannot be discontinued or switched to a different medication before starting study drug.
6. Participants with electrocardiogram (ECG) abnormalities considered by the investigator to be clinically significant, or repeated baseline prolongation of the rate-corrected QT interval (QTc).
7. Ongoing or clinically significant active infection as judged by the investigator.
8. Signs of peripheral neuropathy (PN) ≥ NCI CTCAE Grade 2.
9. Concomitant chemotherapy, hormonal therapy, immunotherapy, or any other form of cancer treatment.
10. Use of strong cytochrome P450 (CYP) 3A4 inhibitors within 2 weeks before the first dose of study drug.
11. Any preexisting medical condition of sufficient severity to prevent full compliance with the study.
12. History of or current neoplasm other than gastric adenocarcinoma, except for curatively treated nonmelanoma skin cancer or in situ carcinoma of the cervix uteri.
13. Known diagnosis of human immunodeficiency virus (HIV) infection (testing is not mandatory).
14. Symptomatic brain metastases.
15. Ongoing anticoagulant therapy (eg, aspirin, coumadin, heparin).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2014-08-04 (Actual); Primary Completion 2016-01-15 (Actual); Study Completion 2016-01-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director Clinical Science, Study Director — Millennium Pharmaceuticals, Inc.
Locations (17):
- United States (7):
  - Aurora, Colorado
  - St. Petersburg, Florida
  - Tampa, Florida
  - Boston, Massachusetts
  - Cincinnati, Ohio
  - Nasheville, Tennessee
  - Nashville, Tennessee
- Belgium (3):
  - Bruges
  - Brussels
  - Leuven
- Spain (4):
  - Barcelona, Barcelona
  - Madrid, Madrid
  - Málaga, Malaga
  - Seville, Sevilla
- United Kingdom (3):
  - London, Greater London
  - Manchester, Greater Manchester
  - Sutton, Surrey

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 24 investigative sites in Belgium, Spain, United Kingdom and the United States from 04 August 2014 to 15 January 2016.
Pre-assignment Details: Participants with a diagnosis of metastatic or recurrent adenocarcinoma of the stomach or gastroesophageal junction expressing Guanylyl Cyclase C (GCC) were enrolled in 1 treatment group, MLN0264 1.8 mg/kg, 30-minute IV infusion, Day 1 of each 21-day cycle.
Groups:
- MLN0264 1.8 mg/kg (GCC Low): MLN0264 1.8 mg/kg, 30-minute intravenous (IV) infusion, Day 1 of each 21-day cycle, for up to 1 year or until disease progression or unacceptable toxicity occurs (Up to 14 cycles). The dose may be decreased, delayed or discontinued in participants who develop treatment-associated nonhematologic and hematologic toxicity to MLN0264. Participants with guanylyl cyclase C (GCC) protein expression=Low (combined H-score 10-59). Total H-score 0-600 is the combined score of cytoplasmic staining 0-300 and apical staining 0-300 and is based on the percentage of tumor cells with staining intensity 1+, 2+ and 3+.
- MLN0264 1.8 mg/kg (GCC Intermediate): MLN0264 1.8 mg/kg, 30-minute IV infusion, Day 1 of each 21-day cycle, for up to 1 year or until disease progression or unacceptable toxicity occurs (Up to 9 cycles). The dose may be decreased, delayed or discontinued in participants who develop treatment-associated nonhematologic and hematologic toxicity to MLN0264. Participants with guanylyl cyclase C (GCC) protein expression=Intermediate (combined H-score 60-119). Total H-score 0-600 is the combined score of cytoplasmic staining 0-300 and apical staining 0-300 and is based on the percentage of tumor cells with staining intensity 1+, 2+ and 3+.
- MLN0264 1.8 mg/kg (GCC High): MLN0264 1.8 mg/kg, 30-minute IV infusion, Day 1 of each 21-day cycle, for up to 1 year or until disease progression or unacceptable toxicity occurs (Up to 8 cycles). The dose may be decreased, delayed or discontinued in participants who develop treatment-associated nonhematologic and hematologic toxicity to MLN0264. Participants with guanylyl cyclase C (GCC) protein expression=Intermediate (combined H-score >120). Total H-score 0-600 is the combined score of cytoplasmic staining 0-300 and apical staining 0-300 and is based on the percentage of tumor cells with staining intensity 1+, 2+ and 3+.
Period: Overall Study
Arm/Group | MLN0264 1.8 mg/kg (GCC Low) | MLN0264 1.8 mg/kg (GCC Intermediate) | MLN0264 1.8 mg/kg (GCC High)
Started | 9 | 15 | 14
Completed | 0 | 0 | 0
Not Completed | 9 | 15 | 14
Not completed — Study Terminated by Sponsor | 3 | 3 | 3
Not completed — Withdrawal by Subject | 2 | 1 | 1
Not completed — Reason not Specified | 4 | 11 | 10

BASELINE CHARACTERISTICS:
Population: Safety population included all participants who received any amount of MLN0264.
Groups:
- Total: Total of all reporting groups
Arm/Group | MLN0264 1.8 mg/kg (GCC Low) | MLN0264 1.8 mg/kg (GCC Intermediate) | MLN0264 1.8 mg/kg (GCC High) | Total
Number analyzed (Participants) | 9 | 15 | 14 | 38
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.1 (7.70) | 62.9 (12.78) | 62.9 (7.86) | 62.2 (9.89)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 5 | 1 | 7
  Male | 8 | 10 | 13 | 31
Race/Ethnicity, Customized [Number; unit: participants]
  Hispanic or Latino | 0 | 0 | 1 | 1
  Not Hispanic or Latino | 9 | 14 | 12 | 35
  Not Reported | 0 | 1 | 1 | 2
Race/Ethnicity, Customized [Number; unit: participants]
  White | 9 | 15 | 12 | 36
  Black or African American | 0 | 0 | 1 | 1
  Asian | 0 | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  Belgium | 1 | 0 | 1 | 2
  United States | 6 | 8 | 8 | 22
  United Kingdom | 0 | 2 | 2 | 4
  Spain | 2 | 5 | 3 | 10
Height [Mean (Standard Deviation); unit: cm] | 169.7 (7.49) | 167.8 (9.85) | 171.1 (9.38) | 169.4 (9.05)
Weight [Mean (Standard Deviation); unit: kg] | 71.51 (11.253) | 71.67 (17.060) | 72.75 (12.597) | 72.03 (13.913)
Body Surface Area [Mean (Standard Deviation); unit: m^2] | 1.832 (0.1683) | 1.818 (0.2520) | 1.854 (0.2014) | 1.835 (0.2113)

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate (ORR) Based on Response Evaluation Criteria in Solid Tumors (RECIST)
Description: ORR is defined as the percentage of participants with complete response (CR) or partial response (PR) as assessed by the investigator using Response Evaluation Criteria In Solid Tumors (RECIST) version 1.1. CR: Disappearance of all target lesions, non-target lesions, no new lesions, and normalization of tumor marker level. PR: At least a 30% decrease in the sum of diameters of target lesions, no progression in non-target lesion, and no new lesions.
Time Frame: Day 21, every other cycle, starting with Cycle 2 until disease progression, death or study closure (up to 17 months)
Population: Response-Evaluable population included all participants with measurable disease who received at least 1 dose of MLN0264 and had at least 1 post-baseline response assessment.
Measure: Number; unit: percentage of participants
Arm/Group | MLN0264 1.8 mg/kg (GCC Low) | MLN0264 1.8 mg/kg (GCC Intermediate) | MLN0264 1.8 mg/kg (GCC High)
Number analyzed (Participants) | 9 | 14 | 13
percentage of participants | 0 | 14 | 0

2. Secondary Outcome: Number of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: An AE is defined as any untoward medical occurrence in a participant administered a pharmaceutical product; the untoward medical occurrence does not necessarily have a causal relationship with this treatment. A serious adverse event (SAE) is defined as any untoward medical occurrence that at any dose results in death, is life-threatening, requires inpatient hospitalization or prolongation of an existing hospitalization, results in persistent or significant disability or incapacity, is a congenital anomaly/birth defect or is a medically important event. Relationship of each AE to study drug will be determined by the Investigator.
Time Frame: From the first dose through 30 days after the last dose of study medication (Up to 10.7 months)
Population: Safety population included all participants who received any amount of MLN0264.
Measure: Number; unit: participants
Arm/Group | MLN0264 1.8 mg/kg (GCC Low) | MLN0264 1.8 mg/kg (GCC Intermediate) | MLN0264 1.8 mg/kg (GCC High)
Number analyzed (Participants) | 9 | 15 | 14
participants
  AEs | 8 | 15 | 14
  SAEs | 2 | 5 | 0

3. Secondary Outcome: Number of Participants With Potentially Clinically Significant Laboratory Evaluation Findings
Description: Participants with at least one post-baseline potentially clinically significant serum chemistry, hematology, coagulation or urinalysis result. Clinically significant results are those that were assessed by the investigator to be Grade 3 or higher using the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE). Grade 3=severe, Grade 4=life threatening or disabling and Grade 5=Death.
Time Frame: From the first dose through 30 days after the last dose of study medication (Up to 10.7 months)
Population: Safety population included all participants who received any amount of MLN0264.
Measure: Number; unit: participants
Arm/Group | MLN0264 1.8 mg/kg
Number analyzed (Participants) | 38
participants
  Chemistry | 8
  Hematology | 13
  Coagulation | 24
  Urinalysis | 0

4. Secondary Outcome: Number of Participants With Potentially Clinically Significant Vital Signs Findings
Description: Participants with at least one potentially clinically significant post-baseline vital sign finding including measurements of diastolic and systolic blood pressure, heart rate, and oral temperature.
Time Frame: Day 1 of each 21 day cycle and 30 days after the last dose of study medication (Up to 10.7 months)
Population: Safety population included all participants who received any amount of MLN0264.
Measure: Number; unit: participants
Arm/Group | MLN0264 1.8 mg/kg
Number analyzed (Participants) | 38
participants | 0

5. Secondary Outcome: Progression Free Survival (PFS)
Description: PFS is defined as the time in days from the date of first study drug administration to the date of first documentation of disease progression or death. Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions.
Time Frame: Time Frame: Day 21 of every other 21-day cycle starting with Cycle 2, 30 days after the last dose of study medication, and then every 12 weeks for up to an additional 6 months (Up to 16.7 months)
Population: as for outcome 1
Measure: Median (Full Range); unit: days
Arm/Group | MLN0264 1.8 mg/kg (GCC Low) | MLN0264 1.8 mg/kg (GCC Intermediate) | MLN0264 1.8 mg/kg (GCC High)
Number analyzed (Participants) | 9 | 14 | 13
days | 40 [38 to 311] | 49 [38 to 316] | 87 [39 to 427]

6. Secondary Outcome: Duration of Response
Description: Duration of response is defined as the time in days from the date of first documentation of a confirmed response to the date of first documentation of disease progression. Per RECIST v1.1 for target lesions and assessed by magnetic resonance imaging (MRI) - CR: Disappearance of all target lesions, non-target lesions, no new lesions, and normalization of tumor marker level. PR: At least a 30% decrease in the sum of diameters of target lesions, no progression in non-target lesion, and no new lesions.
Time Frame: From first documented response until disease progression (Up to 16.7 months)
Population: Participants from the Response-Evaluable population, all participants with measurable disease who received at least 1 dose of MLN0264 and had at least 1 post-baseline response assessment, who had response.
Measure: Median (Full Range); unit: days
Arm/Group | MLN0264 1.8 mg/kg
Number analyzed (Participants) | 2
days | 45.5 [1 to 90]

7. Secondary Outcome: Disease Control Rate
Description: Disease control rate is defined as the percentage of participants with complete response (CR) or partial response (PR) or stable disease (SD) with a minimum of 12 weeks' duration. CR: Disappearance of all target lesions, non-target lesions, no new lesions, and normalization of tumor marker level. PR: At least a 30% decrease in the sum of the Longest Diameter (LD) of target lesions, taking as reference the baseline sum LD and no new lesions. SD: Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for progressive disease (PD) of target lesions, taking as reference the smallest sum LD since the treatment started and no new lesions. Investigator response is based on the Response Evaluation Criteria in Solid Tumors (RECIST) Version 1.1.
Time Frame: Day 21 of every other 21-day cycle starting with Cycle 2, 30 days after the last dose of study medication, and then every 12 weeks for up to an additional 6 months (Up to 16.7 months)
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | MLN0264 1.8 mg/kg (GCC Low) | MLN0264 1.8 mg/kg (GCC Intermediate) | MLN0264 1.8 mg/kg (GCC High)
Number analyzed (Participants) | 9 | 14 | 13
percentage of participants | 11 | 36 | 54

8. Secondary Outcome: Overall Survival (OS)
Description: Overall survival is defined as the time in days from the date of first study drug administration to the date of death.
Time Frame: Until death or 6 months after the last patient completes treatment-whichever occurs first (Up to 17 months)
Population: Response-evaluable population, all participants with measurable disease who received at least 1 dose of MLN0264 and had at least 1 postbaseline response assessment.
Measure: Median (Full Range); unit: days
Arm/Group | MLN0264 1.8 mg/kg (GCC Low) | MLN0264 1.8 mg/kg (GCC Intermediate) | MLN0264 1.8 mg/kg (GCC High)
Number analyzed (Participants) | 9 | 14 | 13
days | 230 [79 to 394] | 156 [49 to 505] | 206 [24 to 427]

9. Secondary Outcome: Cmax: Maximum Observed Serum Concentration for MLN0264
Description: Maximum observed serum concentration (Cmax) is the peak serum concentration of a drug after administration, obtained directly from the serum concentration-time curve.
Time Frame: Cycles 1-3 predose and 10 minutes, 4 hours, and 3, 4, 8 and 15 days postdose. Cycles 4+ predose, 10 minutes, 4 hours, and 4 and 8 days postdose.
Population: Cmax was not a pre-specified secondary outcome measure. No data was collected.
Arm/Group | MLN0264 1.8 mg/kg
Number analyzed (Participants) | 0

10. Secondary Outcome: MLN0264 Serum Concentrations
Description: Blood samples were collected and sent to a laboratory to be tested for serum concentrations of MLN0264.
Time Frame: Cycles 1-3 pre-dose and 10 minutes, 4 hours, and 3, 4, 8 and 15 days post-dose; Cycles 4-9 and 11-14 pre-dose and 10 minutes post-dose; End of Treatment.
Population: Pharmacokinetic (PK)-Evaluable population included all participants who received at least 1 dose of MLN0264 and who had sufficient MLN0264 concentration-time data to permit reliable estimation of MLN0264 exposure. "n" in the categories is the number of participants with data available at the given time-point.
Measure: Mean (Standard Deviation); unit: μg/mL
Arm/Group | MLN0264 1.8 mg/kg
Number analyzed (Participants) | 38
μg/mL
  Cycle 1 Day 1, Pre-Dose (n=37) | 0.0000 (0.00000)
  Cycle 1 Day 1, 10 Minutes Post-Dose (n=37) | 37.0434 (9.93577)
  Cycle 1 Day 1, 4 Hours Post-Dose (n=38) | 26.0047 (6.27538)
  Cycle 1 Day 3, 48 Hours Post-Dose (n=35) | 7.0839 (1.64899)
  Cycle 1 Day 4, 72 Hours Post-Dose (n=35) | 4.4939 (1.25657)
  Cycle 1 Day 8, 168 Hours Post-Dose (n=38) | 1.6795 (0.71586)
  Cycle 1 Day 15, 336 Hours Post-Dose (n=36) | 0.5778 (0.22063)
  Cycle 2 Day 1, Pre-Dose (n=36) | 0.7466 (2.68737)
  Cycle 2 Day 1, 10 Minutes Post-Dose (n=36) | 32.1622 (9.61463)
  Cycle 2 Day 1, 4 Hours Post-Dose (n=36) | 26.0278 (9.43156)
  Cycle 2 Day 3, 48 Hours Post-Dose (n=36) | 7.7186 (2.04169)
  Cycle 2 Day 4, 72 Hours Post-Dose (n=33) | 4.9140 (1.05592)
  Cycle 2 Day 8, 168 Hours Post-Dose (n=35) | 1.7813 (0.49456)
  Cycle 2 Day 15, 336 Hours Post-Dose (n=36) | 0.6959 (0.27579)
  Cycle 3 Day 1, Pre-Dose (n=19) | 0.4905 (0.77805)
  Cycle 3 Day 1, 10 Minutes Post-Dose (n=19) | 31.1505 (8.74114)
  Cycle 3 Day 1, 4 Hours Post-Dose (n=19) | 25.1787 (5.49543)
  Cycle 3 Day 3, 48 Hours Post-Dose (n=14) | 6.7360 (1.56940)
  Cycle 3 Day 4, 72 Hours Post-Dose (n=15) | 5.8887 (3.05461)
  Cycle 3 Day 8, 168 Hours Post-Dose (n=18) | 1.5078 (0.48401)
  Cycle 3 Day 15, 336 Hours Post-Dose (n=18) | 0.6807 (0.25869)
  Cycle 4 Day 1, Pre-Dose (n=16) | 0.3916 (0.16462)
  Cycle 4 Day 1, 10 Minutes Post-Dose (n=15) | 32.3427 (8.33045)
  Cycle 5 Day 1, Pre-Dose (n=7) | 0.4757 (0.18995)
  Cycle 5 Day 1, 10 Minutes Post-Dose (n=7) | 33.9286 (7.14793)
  Cycle 6 Day 1, Pre-Dose (n=8) | 0.4915 (0.34173)
  Cycle 6 Day 1, 10 Minutes Post-Dose (n=8) | 30.3850 (7.79913)
  Cycle 6 Day 4, 72 Hours Post-Dose (n=7) | 5.0676 (1.54862)
  Cycle 6 Day 8, 168 Hours Post-Dose (n=6) | 1.6910 (0.40781)
  Cycle 7 Day 1, Pre-Dose (n=3) | 0.5097 (0.20409)
  Cycle 7 Day 1, 10 Minutes Post-Dose (n=3) | 31.0133 (8.23430)
  Cycle 8 Day 1, Pre-Dose (n=3) | 0.5677 (0.24180)
  Cycle 8 Day 1, 10 Minute Post-Dose (n=3) | 31.6467 (8.93229)
  Cycle 9 Day 1, Pre-Dose (n=2) | 0.9290 (0.49639)
  Cycle 9 Day 1, 10 Minutes Post-Dose (n=2) | 32.3500 (6.77408)
  Cycle 11 Day 1, Pre-Dose (n=1) | 0.7760 (0.00000)
  Cycle 11 Day 1, 10 Minutes Post-Dose (n=1) | 56.8400 (0.00000)
  Cycle 12 Day 1, Pre-Dose (n=1) | 0.7350 (0.00000)
  Cycle 12 Day 1, 10 Minutes Post-Dose (n=1) | 49.8800 (0.00000)
  Cycle 13 Day 1, Pre-Dose (n=1) | 0.8870 (0.00000)
  Cycle 13 Day 1, 10 Minutes Post-Dose (n=1) | 41.6400 (0.00000)
  Cycle 14 Day 1, Pre-Dose (n=1) | 1.0260 (0.00000)
  Cycle 14 Day 1, 10 Minutes Post-Dose (n=1) | 41.9200 (0.00000)
  End of Treatment (n=26) | 0.3323 (0.21216)

11. Secondary Outcome: Serum Concentration of Total Antibodies (Conjugated and Unconjugated)
Description: Blood samples were collected and sent to a laboratory to be tested for conjugated and unconjugated antibodies.
Time Frame: as for outcome 10
Population: PK-Evaluable population included all participants who received at least 1 dose of MLN0264 and who had sufficient MLN0264 concentration-time data to permit reliable estimation of MLN0264 exposure. "n" in the categories is the number of participants with data available at the given time-point.
Measure: Mean (Standard Deviation); unit: μg/mL
Arm/Group | MLN0264 1.8 mg/kg
Number analyzed (Participants) | 38
μg/mL
  Cycle 1 Day 1, Pre-Dose (n=37) | 0.0000 (0.00000)
  Cycle 1 Day 1, 10 Minutes Post-Dose (n=37) | 41.8154 (10.05341)
  Cycle 1 Day 1, 4 Hours Post-Dose (n=38) | 35.7626 (8.46954)
  Cycle 1 Day 3, 48 Hours Post-Dose (n=35) | 16.0664 (3.26969)
  Cycle 1 Day 4, 72 Hours Post-Dose (n=35) | 11.7461 (2.60098)
  Cycle 1 Day 8, 168 Hours Post-Dose (n=38) | 6.1851 (1.73972)
  Cycle 1 Day 15, 336 Hours Post-Dose (n=36) | 3.3926 (1.00149)
  Cycle 2 Day 1, Pre-Dose (n=36) | 2.5995 (3.79916)
  Cycle 2 Day 1, 10 Minutes Post-Dose (n=35) | 43.4749 (9.71796)
  Cycle 2 Day 1, 4 Hours Post-Dose (n=36) | 35.6691 (10.26134)
  Cycle 2 Day 3, 48 Hours Post-Dose (n=36) | 18.4167 (4.07769)
  Cycle 2 Day 4, 72 Hours Post-Dose (n=33) | 13.3398 (3.23987)
  Cycle 2 Day 8, 168 Hours Post-Dose (n=35) | 7.3613 (1.87974)
  Cycle 2 Day 15, 336 Hours Post-Dose (n=36) | 4.3511 (1.47322)
  Cycle 3 Day 1, Pre-Dose (n=19) | 2.5274 (1.54088)
  Cycle 3 Day 1, 10 Minutes Post-Dose (n=19) | 41.3674 (11.88629)
  Cycle 3 Day 1, 4 Hours Post-Dose (n=19) | 33.2692 (9.42530)
  Cycle 3 Day 3, 48 Hours Post-Dose (n=14) | 15.9500 (5.08026)
  Cycle 3 Day 4, 72 Hours Post-Dose (n=15) | 12.8393 (4.56059)
  Cycle 3 Day 8, 168 Hours Post-Dose (n=18) | 7.5035 (2.01984)
  Cycle 3 Day 15, 336 Hours Post-Dose (n=18) | 4.2384 (1.66059)
  Cycle 4 Day 1, Pre-Dose (n=16) | 2.9082 (1.03729)
  Cycle 4 Day 1, 10 Minutes Post-Dose (n=15) | 45.4333 (13.84498)
  Cycle 5 Day 1, Pre-Dose (n=7) | 3.2396 (0.88493)
  Cycle 5 Day 1, 10 Minutes Post-Dose (n=7) | 43.0629 (7.30566)
  Cycle 6 Day 1, Pre-Dose (n=8) | 3.0810 (1.29133)
  Cycle 6 Day 1, 10 Minutes Post-Dose (n=8) | 39.9300 (10.13066)
  Cycle 6 Day 4, 72 Hours Post-Dose (n=7) | 14.7957 (4.09897)
  Cycle 6 Day 8, 168 Hours Post-Dose (n=6) | 9.6217 (1.53148)
  Cycle 7 Day 1, Pre-Dose (n=3) | 3.3417 (1.64015)
  Cycle 7 Day 1, 10 Minutes Post-Dose (n=3) | 42.1667 (8.75528)
  Cycle 8 Day 1, Pre-Dose (n=3) | 3.0573 (1.21148)
  Cycle 8 Day 1, 10 Minute Post-Dose (n=3) | 32.6333 (5.94980)
  Cycle 9 Day 1, Pre-Dose (n=2) | 3.0440 (0.98429)
  Cycle 9 Day 1, 10 Minutes Post-Dose (n=2) | 45.8000 (7.04278)
  Cycle 11 Day 1, Pre-Dose (n=1) | 4.2420 (0.00000)
  Cycle 11 Day 1, 10 Minutes Post-Dose (n=1) | 44.3000 (0.00000)
  Cycle 12 Day 1, Pre-Dose (n=1) | 4.1020 (0.00000)
  Cycle 12 Day 1, 10 Minutes Post-Dose (n=1) | 47.3800 (0.00000)
  Cycle 13 Day 1, Pre-Dose (n=1) | 4.9900 (0.00000)
  Cycle 13 Day 1, 10 Minutes Post-Dose (n=1) | 55.2600 (0.00000)
  Cycle 14 Day 1, Pre-Dose (n=1) | 5.6750 (0.00000)
  Cycle 14 Day 1, 10 Minutes Post-Dose (n=1) | 61.5000 (0.00000)
  End of Treatment (n=26) | 2.5393 (1.32302)

12. Secondary Outcome: Serum Concentration of Monomethyl Auristatin E (MMAE)
Description: Blood samples were collected and sent to a laboratory to be tested for MMAE.
Time Frame: as for outcome 10
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | MLN0264 1.8 mg/kg
Number analyzed (Participants) | 38
ng/mL
  Cycle 1 Day 1, Pre-Dose (n=37) | 0.000 (0.0000)
  Cycle 1 Day 1, 10 Minutes Post-Dose (n=37) | 0.473 (0.6503)
  Cycle 1 Day 1, 4 Hours Post-Dose (n=38) | 2.659 (1.5489)
  Cycle 1 Day 3, 48 Hours Post-Dose (n=35) | 6.153 (3.2773)
  Cycle 1 Day 4, 72 Hours Post-Dose (n=35) | 5.856 (3.4519)
  Cycle 1 Day 8, 168 Hours Post-Dose (n=38) | 2.945 (1.8899)
  Cycle 1 Day 15, 336 Hours Post-Dose (n=36) | 0.532 (0.6693)
  Cycle 2 Day 1, Pre-Dose (n=36) | 0.116 (0.1118)
  Cycle 2 Day 1, 10 Minutes Post-Dose (n=35) | 0.425 (0.2697)
  Cycle 2 Day 1, 4 Hours Post-Dose (n=36) | 2.665 (1.7137)
  Cycle 2 Day 3, 48 Hours Post-Dose (n=36) | 6.746 (4.2361)
  Cycle 2 Day 4, 72 Hours Post-Dose (n=33) | 6.111 (3.6283)
  Cycle 2 Day 8, 168 Hours Post-Dose (n=35) | 2.898 (2.2974)
  Cycle 2 Day 15, 336 Hours Post-Dose (n=36) | 0.579 (0.6221)
  Cycle 3 Day 1, Pre-Dose (n=19) | 0.094 (0.1240)
  Cycle 3 Day 1, 10 Minutes Post-Dose (n=18) | 0.428 (0.4487)
  Cycle 3 Day 1, 4 Hours Post-Dose (n=19) | 2.302 (1.8893)
  Cycle 3 Day 3, 48 Hours Post-Dose (n=14) | 4.493 (2.6877)
  Cycle 3 Day 4, 72 Hours Post-Dose (n=15) | 3.638 (1.8570)
  Cycle 3 Day 8, 168 Hours Post-Dose (n=18) | 2.135 (1.7030)
  Cycle 3 Day 15, 336 Hours Post-Dose (n=17) | 0.342 (0.3637)
  Cycle 4 Day 1, Pre-Dose (n=16) | 0.081 (0.0865)
  Cycle 4 Day 1, 10 Minutes Post-Dose (n=15) | 0.304 (0.1781)
  Cycle 5 Day 1, Pre-Dose (n=7) | 0.084 (0.0331)
  Cycle 5 Day 1, 10 Minutes Post-Dose (n=7) | 0.278 (0.1325)
  Cycle 6 Day 1, Pre-Dose (n=8) | 0.093 (0.0654)
  Cycle 6 Day 1, 10 Minutes Post-Dose (n=7) | 0.322 (0.2232)
  Cycle 6 Day 4, 72 Hours Post-Dose (n=7) | 6.183 (3.3587)
  Cycle 6 Day 8, 168 Hours Post-Dose (n=6) | 2.417 (1.6379)
  Cycle 7 Day 1, Pre-Dose (n=3) | 0.044 (0.0083)
  Cycle 7 Day 1, 10 Minutes Post-Dose (n=3) | 0.115 (0.0439)
  Cycle 8 Day 1, Pre-Dose (n=3) | 0.058 (0.0103)
  Cycle 8 Day 1, 10 Minute Post-Dose (n=3) | 0.132 (0.0425)
  Cycle 9 Day 1, Pre-Dose (n=2) | 0.021 (0.0291)
  Cycle 9 Day 1, 10 Minutes Post-Dose (n=2) | 0.158 (0.0721)
  Cycle 11 Day 1, Pre-Dose (n=1) | 0.093 (0.0000)
  Cycle 11 Day 1, 10 Minutes Post-Dose (n=1) | 0.186 (0.0000)
  Cycle 12 Day 1, Pre-Dose (n=1) | 0.087 (0.0000)
  Cycle 12 Day 1, 10 Minutes Post-Dose (n=1) | 0.167 (0.0000)
  Cycle 13 Day 1, Pre-Dose (n=1) | 0.074 (0.0000)
  Cycle 13 Day 1, 10 Minutes Post-Dose (n=1) | 0.132 (0.0000)
  Cycle 14 Day 1, Pre-Dose (n=1) | 0.081 (0.0000)
  Cycle 14 Day 1, 10 Minutes Post-Dose (n=1) | 0.165 (0.0000)
  End of Treatment (n=25) | 0.173 (0.3359)

13. Secondary Outcome: Number of Participants With Reduction From Baseline in Tumor Size
Description: The number of participants with the best percentage of tumor reduction from baseline in the sum of the diameter was calculated.
Time Frame: as for outcome 7
Population: Response-Evaluable Population was defined as all participants with measurable disease who receive at least 1 dose of MLN0264 and have at least 1 postbaseline response assessment.
Measure: Number; unit: participants
Arm/Group | MLN0264 1.8 mg/kg (GCC Low) | MLN0264 1.8 mg/kg (GCC Intermediate) | MLN0264 1.8 mg/kg (GCC High)
Number analyzed (Participants) | 9 | 14 | 13
participants | 1 [38 to 311] | 2 [38 to 316] | 4 [42 to 427]

14. Secondary Outcome: Guanylyl Cyclase C (GCC) H-score Assessed by Immunohistochemistry (IHC)
Description: Analysis of GCC protein expression levels in tumor tissue (fresh biopsy pretreatment and whenever a biopsy is considered medically safe and technically feasible) was performed using a semiquantitative immunohistochemistry (IHC) assay and the total GCC H-Score was determined. GCC H-score is based on the sum of the 0 to 300 H-score for cytoplasmic staining and the 0 to 300 H-score for apical staining for a total possible H-score 0 to 600. Separate consent was required to obtain archival tumor specimens for GCC expression assessment prior to screening.
Time Frame: Approximately 20 months
Population: Safety population included all participants who received any amount of MLN0264.
Measure: Mean (Full Range); unit: scores on a scale
Arm/Group | MLN0264 1.8 mg/kg (GCC Low) | MLN0264 1.8 mg/kg (GCC Intermediate) | MLN0264 1.8 mg/kg (GCC High)
Number analyzed (Participants) | 9 | 15 | 14
scores on a scale | 74.8 [27 to 100] | 154.6 [110 to 230] | 344.3 [260 to 480]

15. Secondary Outcome: Number of Participants With Antitherapeutic Antibodies (ATA)
Description: Blood samples were collected to assess the immunogenicity of MLN0264 (ATA development) using a laboratory test. Neutralizing ATA assessment was performed for ATA-positive samples only.
Time Frame: Pre-dose of each 21 day cycle and 30 days after last dose of study medication (Up to 10.7 months)
Population: Safety Population included all participant who received any amount of MLN0264.
Measure: Number; unit: participants
Arm/Group | MLN0264 1.8 mg/kg (GCC Low) | MLN0264 1.8 mg/kg (GCC Intermediate) | MLN0264 1.8 mg/kg (GCC High)
Number analyzed (Participants) | 9 | 15 | 14
participants | 0 | 3 | 1

ADVERSE EVENTS:
Time Frame: From the first dose through 30 days after the last dose of study drug (up to 10.7 Months)
Description: At each visit the investigator documented any occurrence of AEs and abnormal laboratory findings. Any event spontaneously reported by participant or observed by investigator was recorded, irrespective of relation to study treatment.
Arm/Group | MLN0264 1.8 mg/kg
Serious Adverse Events (participants affected / at risk) | 7/38
Other Adverse Events (participants affected / at risk) | 37/38
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | MLN0264 1.8 mg/kg (N=38)
Diarrhoea (Gastrointestinal disorders) | 1
Dysphagia (Gastrointestinal disorders) | 1
Upper gastrointestinal hemorrhage (Gastrointestinal disorders) | 1
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 — One treatment-emergent death occurred during treatment with MLN0264 with and is not related.
Tumour hemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Anaemia (Blood and lymphatic system disorders) | 1
Supraventricular tachycardia (Cardiac disorders) | 1
Bile duct obstruction (Hepatobiliary disorders) | 1
Hip fracture (Injury, poisoning and procedural complications) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | MLN0264 1.8 mg/kg (N=38)
Anaemia (Blood and lymphatic system disorders) | 6
Neutropenia (Blood and lymphatic system disorders) | 5
Abdominal pain (Gastrointestinal disorders) | 4
Ascites (Gastrointestinal disorders) | 2
Constipation (Gastrointestinal disorders) | 9
Diarrhoea (Gastrointestinal disorders) | 6
Dysphagia (Gastrointestinal disorders) | 3
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 2
Nausea (Gastrointestinal disorders) | 20
Stomatitis (Gastrointestinal disorders) | 3
Vomiting (Gastrointestinal disorders) | 10
Asthenia (General disorders) | 10
Fatigue (General disorders) | 12
Oedema peripheral (General disorders) | 7
Pain (General disorders) | 2
Pyrexia (General disorders) | 4
Urinary tract infection (Infections and infestations) | 2
Fall (Injury, poisoning and procedural complications) | 2
Blood alkaline phosphatase increased (Investigations) | 4
Gamma-glutamyltransferase increased (Investigations) | 4
Neutrophil count decreased (Investigations) | 4
Weight decreased (Investigations) | 3
Decreased appetite (Metabolism and nutrition disorders) | 11
Dehydration (Metabolism and nutrition disorders) | 3
Hyperglycaemia (Metabolism and nutrition disorders) | 3
Hypoalbuminaemia (Metabolism and nutrition disorders) | 4
Hypocalcaemia (Metabolism and nutrition disorders) | 4
Hypokalaemia (Metabolism and nutrition disorders) | 2
Hypomagnesaemia (Metabolism and nutrition disorders) | 2
Hyponatraemia (Metabolism and nutrition disorders) | 2
Back pain (Musculoskeletal and connective tissue disorders) | 4
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 3
Myalgia (Musculoskeletal and connective tissue disorders) | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4
Dizziness (Nervous system disorders) | 2
Hypoaesthesia (Nervous system disorders) | 2
Neuropathy peripheral (Nervous system disorders) | 4
Tremor (Nervous system disorders) | 2
Confusional state (Psychiatric disorders) | 2
Depression (Psychiatric disorders) | 2
Proteinuria (Renal and urinary disorders) | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4
Orthopnoea (Respiratory, thoracic and mediastinal disorders) | 2
Alopecia (Skin and subcutaneous tissue disorders) | 5
Deep vein thrombosis (Vascular disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
In general, Investigators may publish clinical data after the earlier of (i) publication by the Sponsor or (ii) 12 months following the abandonment, early termination or database lock; provided a copy of the publication provided to Sponsor at least 30 days ahead of publication, the Sponsor's confidential information is removed as may be requested by Sponsor and Investigator defers publication for up to 60 days in the event Sponsor provides notice that it intends to file a patent application.